CLINICAL TRIAL: NCT07261514
Title: Correlation Between Triglyceride Glucose Index and Myocardial Infarct Size, Microcirculation Obstruction and Intramyocardial Hemorrhage in Patients With ST-segment Elevation Myocardial Infarction.
Brief Title: Correlation Between Triglyceride Glucose Index and Myocardial Injury Assessed by Cardiac Magnetic Resonance Imaging (CMR) in Patients With STEMI
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Anzhen Hospital (Other); Beijing Chao Yang Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); First People's Hospital of Yulin (Other); Wuhan Asia Heart Hospital (Other); Zunyi Medical College (Other)
Responsible Party: Principal Investigator, Qian geng, Associate Chief Physician, Chinese PLA General Hospital
Other Study IDs: 2025QG-TyG index
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2014-01

CONDITIONS: ST Elevation (STEMI) Myocardial Infarction
Keywords: ST-segment elevation Myocardial Infarction; triglyceride glucose index; Cardiac magnetic resonance; myocardial infarct size; intramyocardial hemorrhage; microvascular obstruction
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- low TyG index group: Patients with a TyG index below 1.41 were categorized into the low TyG group.
- medium TyG index: Patients with a TyG index between 1.41 and 1.96 were categorized into the medium TyG group.
- high TyG index group: Patients with a TyG index greater than 1.96 were categorized into the high TyG index group.

SUMMARY:
This research aim is to investigate the correlation between triglyceride glucose index (TyG index) and myocardial infarct size, microcirculation obstruction (MVO) and intramyocardial hemorrhage (IMH) assessed by cardiac magnetic resonance imaging (CMR) in patients with ST-segment elevation myocardial infarction (STEMI), and to evaluate its value as a potential predictor of myocardial injury.To further determine the influence of TyG index on the prognosis of STEMI patients after PCI.This cohort included 674 patients with STEMI undergoing primary percutaneous coronary intervention (pPCI). Baseline clinical data were collected and cardiac magnetic resonance imaging was performed approximately 7 days after Acute Myocardial Infarction(AMI). Patients were divided into three groups according to the TyG index , namely high TyG index group, medium TyG index group and low TyG index group. Multiple linear regression, Pearson/Spearman correlation analysis and Logistics regression analysis were used to analyze the correlation between TyG index and myocardial infarct size, microcirculation obstruction and intramyocardial hemorrhage.Eventually, we came to the conclusion that the TyG index was independently associated with severity of myocardial injury after STEMI as assessed by CMR. TyG index is not only an independent predictor of microcirculation disturbance in STEMI patients, but also significantly correlated with poor cardiovascular prognosis. is a powerful marker for stratifying risk of adverse cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* 1) patients meet diagnostic criteria for STEMI-"The priority for these patients is the implementation of reperfusion therapy as soon as possible .In the appropriate clinical context,ST-segment elevation (accessed at the J-point) indicates possible acute coronary artery in the following situations:New ST elevation at the J-point in at least two contiguous leads:·≥ 2.5 mm in men under 40years,≥2mm in males 40 years and older,or ≥1.5mmin women relatively less of age in leads V2-V3,and/or ≥1mm in the other leads (in the absence of left ventricular hypertrophy or left bundle branch block) Post-STEMI reperfusion with PCI, diagnosis and treatment strategy in accordance with current diagnosis and treatment standards and guidelines27" and complete pPCI within 48h-"" diagnostic strategy meets current diagnostic criteria and guidelines;2) KillIP<3 and consent to CMR examination and follow-up observation, and CMR examination is completed within 7 days after surgery. 3) Monitor baseline blood glucose and baseline triglycerides during admission.

Exclusion criteria: 1) Patients with NSTEMI 2) Lack of clinical data 3) Presence of contraindications to CMR examination-such as implantable cardiac pacemaker, clo gadolinium contrast agent or renal insufficiency; meanwhile, patients with Killip IV cardiac function or clinical instability, and patients with valvular disease, congenital heart disease, pulmonary hypertension, cardiomyopathy history, persistent atrial fibrillation, etc. affecting cardiac structure and function parameters were excluded; Patients with previous history of myocardial infarction, coronary artery intervention and coronary artery bypass grafting were also excluded; patients with severe clinical diseases such as severe hematological diseases, infectious diseases, malignant tumors, liver and kidney failure, and mental disorders or intellectual disabilities who could not cooperate with examination and follow-up; 4) patients with poor MRI quality or sequence deletion were not included in the study.

Exclusion Criteria:

* Contraindications of CMR examination, such as implantable cardiac pacemaker, claustrophobia, allergy to gadolinium contrast agent or renal insufficiency; meanwhile, patients with Killip IV cardiac function or unstable clinical condition, as well as patients with valve disease, congenital heart disease, pulmonary hypertension, cardiomyopathy history, persistent atrial fibrillation, etc. affecting cardiac structure and function parameters shall be excluded; Patients with a history of myocardial infarction, coronary artery intervention, or coronary artery bypass grafting were also excluded. Patients with severe hematological diseases, infectious diseases, malignant tumors, liver and kidney failure, mental disorders or intellectual disabilities who could not cooperate with examination and follow-up, or poor or missing MRI images were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary PCI-treated patients with acute STEMI
Sampling Method: Probability Sample
Enrollment: 674 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
major adverse cardiovascular events | 4 years after discharge
  Death , recurrence of myocardial infarction, heart failure after discharge

SECONDARY OUTCOMES:
myocardial infarct size | Cardiac MRI within 7 days after surgery
  LGE sequences are acquired from CMR .The LGE images were analyzed manually or semi-automatically with software tools to calculate the size or volume of the infarct area .
Microvascular occlusion | Cardiac MRI within 7 days after surgery
  T1-weighted sequences are acquired from CMR and analyzed by software.Identified by early or late gadolinium-enhanced imaging using T1-weighted sequences with high inversion times
Intramyocardial hemorrhage (IMH) | Cardiac MRI within 7 days after surgery
  IMH was detected by T2-weighted imaging or T2 mapping, identified using low signal areas.

CONTACTS AND LOCATIONS:
Overall Officials: geng qian, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China